CLINICAL TRIAL: NCT04682340
Title: Analysis of Bisphenol A Concentration in Serum in Women of Reproductive Age With Autoimmune Thyroid Disease
Brief Title: Analysis of BPA Concentration in Serum in Women of Reproductive Age With Autoimmune Thyroid Disease
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Karolina Zawadzka, Principal Investigator, Jagiellonian University
Other Study IDs: BPA-Thyroid
Record Dates: First submitted 2020-12-13; First posted 2020-12-23 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Hypothyroidism; Hyperthyroidism; Hashimoto Disease; Graves Disease
Keywords: bisphenol A; BPA; Hashimoto's Disease; Graves' Disease
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism; Hashimoto Disease; Graves Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hashimoto's Group: Thyroid antibody positive and hypothyroidism
  Interventions: Diagnostic Test: Serum BPA
- Graves' Group: Thyroid antibody positive and hyperthyroidism
  Interventions: Diagnostic Test: Serum BPA
- Control Group: Thyroid antibody negative and euthyroidism
  Interventions: Diagnostic Test: Serum BPA

INTERVENTIONS:
Diagnostic Test: Serum BPA — Serum BPA levels will be compared between women with autoimmune thyroid disease and normal women.

SUMMARY:
The aim of the study is to assess the relationship between the concentration of bisphenol A in serum and selected parameters of thyroid function in women of reproductive age with thyroid dysfunction - Hashimoto's disease and Graves' disease.

ELIGIBILITY:
Inclusion Criteria:

* Graves' disease or Hashimoto's disease (positive thyroid autoantibody)
* Control group: thyroid autoantibody negative, normal thyroid function
* Women aged 18 to 45 in both the control group and experimental group

Exclusion Criteria:

* Pregnancy and lactating women
* Previous or planned treatment with 131I or thyroidectomy
* The use of drugs affecting the thyroid function (lithium, amiodarone, interferon a, sodium nitroprusside, sunitinib, sorafenib, iodine contrast, antibiotics / antifungals / antivirals (for at least 4 weeks prior to recruitment to the study), which do not result from the treatment of thyroid disease (levothyroxine, thyreostatic drugs, glucocorticoids)
* Active malignancy
* Other autoimmune diseases
* Other endocrine diseases
* Patients with severe liver, kidney or heart failure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women in the reproductive age from 18 to 45 years of age will be qualified to the study group. Women will be recruited from among patients admitted to the University Hospital in Krakow. After qualifying for the study, each patient will be collected demographic data, information about medical history and medications, as well as anthropometric data.During the medical visit, patients will be presented with all information about participation in the study and only those who give their informed consent in writing will be qualified for the study. Based on the clinical picture and the results of laboratory tests (the level of TSH, fT4 in the plasma and the presence of thyroid autoantibodies), the patients will be divided into 2 groups - 30 women with hyperthyroidism, 30 women with hypothyroidism. 20 healthy women without any thyroid dysfunction will be the control group. The groups will be matched according to age, body mass index and smoking.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Comparison of serum BPA levels between the group with AITD and control group | Dec 2020 - April 2021

SECONDARY OUTCOMES:
The association between serum BPA levels and serum thyroid hormone levels in the AITD group | Dec 2020 - April 2021
  To determine the association between serum BPA concentrations and serum thyroid hormone levels in adult women

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Medical College, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: No